CLINICAL TRIAL: NCT01559974
Title: Phase 4 Study of 25-hydroxy-vitamin D in Patients With Peripheral Artery Occlusive Disease and Walking Ability
Brief Title: Vitamin D and Walking Ability in Patients With Peripheral Artery Occlusive Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P Vit D 23032011 v2
Record Dates: First submitted 2011-12-01; First posted 2012-03-21 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral arterial disease; PAOD; Vitamin D; Walking impairment
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Active Comparator)
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo to 45'000 units of Cholecalciferol per month for 3 months
  Arms: Placebo
Drug: Cholecalciferol — 45'000 units of cholecalciferol per month for 3 months
  Arms: Vitamin D

SUMMARY:
The purpose of this study is to determine whether the intake of Vitamin D has a positive effect on walking ability of patients with peripheral artery occlusive disease. Skeletal muscle fibers change morphology in peripheral artery occlusive disease. In patients with Vitamin D-deficiency there are also changes of skeletal muscle fibers. The investigators have the hypothesis that patients with peripheral artery occlusive disease with subsequent changes of muscle fibers morphology of calf muscles might take profit of the administration of Vitamin D in combination with training.

DETAILED DESCRIPTION:
Background On the one hand, patients suffering from peripheral artery occlusive disease may have a significant decrease in their walking ability. When there is insufficient supply of oxygen to the muscles, especially the calf muscles, structural changes of skeletal muscle fibers appear. On the other hand, these patients might also have an insufficient supply with Vitamin D as it is often the case in the general population. A deficiency of Vitamin D also causes structural changes in the skeletal muscles and causes muscle weakness.

Hypothesis Vitamin D - intake can improve the walking ability of patients with peripheral artery occlusive disease and eventually Vitamin D - deficiency.

Aim of the study To evaluate the influence of Vitamin D - intake on walking ability of patients with peripheral artery occlusive disease, which would be a simple, safe and non-invasive measure with a positive effect on quality of life and indirectly on cardiovascular health in general (better mobility).

Primary endpoint:

Measurement of walking ability with treadmill test at the beginning and after a 3 month-treatment with Vitamin D, in combination with a home-based training.

Secondary endpoints:

* Measurement of calf muscle perfusion as an indirect parameter for walking ability, measurement at the beginning, after three months and after a 6 month follow up.
* Quality of life questionnaires (SF 36 and walking impairment questionnaire), visual analogue scale.

Study design:

Prospective, randomised, double-blind, placebo-controlled, investigator-initiated pilot study with a study duration of 3 months and a 3 month - follow up.

Study course:

6 study visits are planned.

* Visit 0: screening visit, lab (Calcium, Vitamin D3), questionnaires
* Visit 1: treadmill test, measurement of calf muscle perfusion, intake of first monthly dose of Cholecalciferol 45'000 units (or placebo)
* Visit 2 (after 1 month): vital parameters, second dose of 45'000 units of Cholecalciferol (or placebo)
* Visit 3 (after 2 months): vital parameters, third dose of 45'000 units of Cholecalciferol (or placebo)
* Visit 4 (after 3 months): treadmill test, measurement of calf muscle perfusion , lab (Calcium, Vitamin D3), questionnaires
* Visit 5 (after 6 months): treadmill test, measurement of calf muscle perfusion , lab (Calcium, Vitamin D3), questionnaires

ELIGIBILITY:
Inclusion Criteria:

* peripheral artery obliterative disease Rutherford 1 to 3
* informed consent
* motivation

Exclusion Criteria:

* inability of treadmill walking
* not motivated
* female patients: childbearing age (age limit 49 years)
* PTA or surgical revascularisation within 3 months before study entry
* cancer, life expectancy lower than 6 months
* ongoing therapy with Vitamin D
* 25-OH-Vitamin D level 125 nmol/l and above
* contraindications for Vitamin D intake (sarcoidosis, acute lung tbc, hypercalcemia, intake of Vitamin D analogs
* contraindications for ultrasound contrast agent (known hypersensitivity, recent acute coronary syndrome, unstable ischemic heart disease, after PTCA, heart insufficiency NYHA III or IV, severe rhythm disorders, known right- left shunt, severe pulmonary artery hypertension, adult respiratory distress syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline initial claudication distance (ICD) at 3 months | 3 months
  Follow up after 6 months.
Change from baseline absolute claudication distance (ACD) at 3 months | 3 months
  Follow up after 6 months.

SECONDARY OUTCOMES:
Change from baseline Vitamin D3 at 3 months | 3 months
  Follow up after 6 months.
Change of baseline Calcium at 3 months | 3 months
  Follow up after 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt A Jaeger, Prof, Principal Investigator — University of Basel
Locations (1):
- University Hospital, Basel, Canton of Basel-City, Switzerland